CLINICAL TRIAL: NCT03168789
Title: Smartphone Delivered Meditation for BP Control Among Prehypertensives
Brief Title: Tension Tamer Randomized Control Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Responsible Party: Principal Investigator, Frank Treiber, Professor and Director TACHL, College of Nursing, Medical University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00020894
Record Dates: First submitted 2017-05-25; First posted 2017-05-30 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Pre-hypertension
Keywords: Breathing Awareness Meditation,
MeSH Terms: conditions — Prehypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tension Tamer (TT) (Experimental): Breathing Awareness Mediation delivered by smartphone app.
  Interventions: Behavioral: Tension Tamer (TT)
- Lifestyle education program (SPCTL) (Active Comparator): Healthy lifestyle education provided by text messages and links to media. Runkeeper app to log physical activity.
  Interventions: Behavioral: Lifestyle education program (SPCTL)

INTERVENTIONS:
Behavioral: Tension Tamer (TT) — Tension Tamer is an app that provides training and motivation for breathing awareness meditation (BAM). The app also tracks heart rate values during each session by placing a finger tip over the rear camera.
  Arms: Tension Tamer (TT)
Behavioral: Lifestyle education program (SPCTL) — SPCTL group will use Runkeeper app to log physical activity. They will also receive text messages with short healthy lifestyle tips, and links to media with pamphlets or videos with more in-depth information.
  Arms: Lifestyle education program (SPCTL)

SUMMARY:
This study is 12 months long and consists of 5 visits at baseline, months 1, 3, 6, and 12. To determine eligibility potential subjects will have resting blood pressures (BP) measured on 2 occasions. Pre-hypertensive individuals will be invited to participate in the study. After informed consent is obtained, subjects will complete baseline visit consisting of a survey, resting BP, wear activity watch for 7 days ambulatory blood pressure monitor for 24-hours, collect saliva and urine samples. Subjects will then be randomly assigned to Tension Tamer (TT) or lifestyle education program delivered via smartphone (SPCTL) groups. At the remaining 4 visits subjects will again complete a survey, resting BP, wear activity watch for 7 days ambulatory blood pressure monitor for 24-hours, collect saliva and urine samples. Throughout the 12 months TT group will meditate twice daily and SPCTL group will log physical activity.

DETAILED DESCRIPTION:
80 stage 1 or 2 pre-hypertensive adults, will be randomly assigned to 2x daily TT at scheduled decreasing doses or enhanced standard of care lifestyle education program delivered via smartphone (SPCTL) for 12 months. Subjects will participate in 5 study visits at baseline/enrollment, 1, 3, 6 , and 12 months

TT subjects will be given the TT app. The app provides instructions on breathing awareness meditation (BAM): focusing upon the moment by sustaining one's attention upon diaphragm movements and related sensations while breathing in a slow, deep, relaxed manner. One learns to passively observe thoughts, images and extraneous sounds without making judgments about them. BAM doesn't involve analysis of historical or recent stressful experiences, but instead centers upon learning to stay in the present moment while meditating. The app will also collect heart rate (HR) values during each session using the phone's camera. The duration of the TT sessions will begin at 15 min., decrease to 10 min., and finally decrease to 5 min. Adherence will be monitored by the receipt of date-stamped heart rate values collected during each meditation session.

SPCTL subjects will be provided Runkeeper app and taught how to record physical activity they perform. Recommended dosage of using SPCTL media and/or app will be that of the TT group. Adherence to SPCTL will be assessed using server file analyses of modules used and activity recorded in Runkeeper.

ELIGIBILITY:
Inclusion Criteria:

1. 18-90 years old, male or female, African American (AA) or White;
2. Stage 1 or 2 pre-hypertensive (i.e., SBP 120-139/DBP<90) based upon 2 consecutive clinic evaluations;
3. Body Mass Index (BMI) 18.5 -45 Kg/m2;
4. legally competent;
5. able to use a smart phone.

Exclusion Criteria:

1. failure to meet any inclusion criteria;
2. type two diabetes or chronic kidney disease (GFR<50 mL/1.7 m2/min.);
3. cancer diagnosis or treatment in past 2 years;
4. prior cardiovascular event, congestive heart failure or angina;
5. prior or current psychiatric illness;
6. ongoing substance abuse (e.g., >21 drinks/week);
7. pharmacologic medications which may influence blood pressure (BP);
8. planned pregnancy;
9. vulnerable populations such as pregnant or nursing women, prisoners, and institutionalized individuals.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2019-11-22 (Actual); Study Completion 2019-11-22 (Actual)

PRIMARY OUTCOMES:
Resting BP | 12 months
  Resting SBP reduction target -7 mmHg.

SECONDARY OUTCOMES:
Ambulatory SBP | 12 months
  24-hr SBP reduction target -4 mmHg.

CONTACTS AND LOCATIONS:
Overall Officials: Frank A Treiber, PhD, Principal Investigator — MUSC College of Nursing
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Adams ZW, Sieverdes JC, Brunner-Jackson B, Mueller M, Chandler J, Diaz V, Patel S, Sox LR, Wilder S, Treiber FA. Meditation smartphone application effects on prehypertensive adults' blood pressure: Dose-response feasibility trial. Health Psychol. 2018 Sep;37(9):850-860. doi: 10.1037/hea0000584. Epub 2018 Jul 16. PMID 30010353